CLINICAL TRIAL: NCT06140667
Title: Comparative Evaluation of the Laryseal TM Pro Laryngeal Mask Airway With Ambu Aura Gain Laryngeal Mask Airway in Anesthetized Paralyzed Adult Patients Undergoing Elective Ophthalmological Surgeries. A Randomized Controlled Study
Brief Title: Laryseal Pro LMA Versus Ambu Aura Gain LMA in Elective Ophthalmological Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Abdelhaleem Abdelrahman, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MK-2023
Record Dates: First submitted 2023-10-31; First posted 2023-11-20 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Laryngeal Masks Comparison

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LarysealTM Pro (Other)
  Interventions: Device: Ambu Aura Gain
- Ambu Aura Gain (Other)
  Interventions: Device: LarysealTM Pro

INTERVENTIONS:
Device: LarysealTM Pro — The LarysealTM Pro is the new generation mask for safe and effective airway management, as it could reduce the risk of aspiration by the integrated suction catheter port to allow effective removal of fluids and gastric contents. So that, it could be a promising airway device as its symmetrical cuff and tube contoured to match the oropharyngeal anatomy for quick and easy first time insertion success. It could be applied in both routine and advanced airway management for patients with a higher risk of a difficult airway, unexpected intubation difficulties, beside to airway control during anesthesia. It was presented in the clinical market in sizes 3, 4 and 5 (according to the body weight; size 3: 30-50Kg, size 4: 50-70 Kg, and size 5:70-100Kg) that can accept larger tracheal tube up to 7.5 and 8mm inner diameter respectively with maximum suction catheter size of 16 Fr.
  Arms: Ambu Aura Gain
Device: Ambu Aura Gain — The AuraGain is Ambu ꞌs 3rd generation disposable laryngeal mask, satisfying 3 fundamental airway management needs by integrating gastric access channel for managing gastric content and intubation capability using standard ET-tubes in an anatomically curved single-use device that facilitates rapid establishment of a safe airway through integrated bite absorption area that could prevent airway occlusion. Other characters include pilot balloon that identifies mask size and provides tactile indication of degree of inflation, navigation marks for guiding flexible scope and is made of phthalate-free material. Its thin and soft cuff is designed to deliver high seal pressure up to 40 cmH2O. It was presented in the clinical market in sizes 3, 4, 5 and 6 (according to the body weight; size 3: 30-50 kg, size 4: 50-70 kg, size 5: 70-100 kg, and size 6: >100 kg) with maximum suction catheter size of 16 Fr.
  Arms: LarysealTM Pro

SUMMARY:
Tracheal intubation is considered the gold standard for protecting the airway. As the supraglottic airway devices (SADs) could be inserted without laryngoscopy, so that SADs with different designs and safety issues could be used to manage difficult airways in anesthesia and emergency medicine with continuous patient oxygenation &ventilation, less hemodynamic stress response and less postoperative complications. Many health care providers do not have the requisite knowledge and enough practice to perform safe and quick intubation. For these providers, SADs can be a valid alterative especially in untrained personnel, or when tracheal intubation is impossibe.

Both devices are with a cuff modified to improve the seal around the glottis and a drainage tube to provide a bypass channel for regurgitated gastric contents, prevent gastric insufflation, and allow the passage of a gastric tube. These features are designed to improve the safety of the mask and broaden its scope, especially when used with positive pressure ventilation.

The AuraGain is Ambu ꞌs 3rd generation disposable laryngeal mask, satisfying 3 fundamental airway management needs by integrating gastric access channel for managing gastric content and intubation capability using standard ET-tubes in an anatomically curved single-use device that facilitates rapid establishment of a safe airway through integrated bite absorption area that could prevent airway occlusion. Other characters include pilot balloon that identifies mask size and provides tactile indication of degree of inflation, navigation marks for guiding flexible scope and is made of phthalate-free material. Its thin and soft cuff is designed to deliver high seal pressure up to 40 cmH2O. It was presented in the clinical market in sizes 3, 4, 5 and 6 (according to the body weight; size 3: 30-50 kg, size 4: 50-70 kg, size 5: 70-100 kg, and size 6: >100 kg) that can accept tracheal tube in sizes ranging from 6.5 up to 7.5 and 8mm inner diameter respectively with maximum suction catheter size of 16 Fr.

The LarysealTM Pro is the new generation mask for safe and effective airway management, as it could reduce the risk of aspiration by the integrated suction catheter port to allow effective removal of fluids and gastric contents. So that, it could be a promising airway device as its symmetrical cuff and tube contoured to match the oropharyngeal anatomy for quick and easy first time insertion success. It could be applied in both routine and advanced airway management for patients with a higher risk of a difficult airway, unexpected intubation difficulties, beside to airway control during anesthesia. It was presented in the clinical market in sizes 3, 4 and 5 (according to the body weight; size 3: 30-50Kg, size 4: 50-70 Kg, and size 5:70-100Kg) that can accept larger tracheal tube up to 7.5 and 8mm inner diameter respectively with maximum suction catheter size of 16 Fr. The Laryseal pro could provide a rapid and secure airway management and improve patient safety with gastric access reducing the risk of pulmonary aspiration, in addition to speeding up the ETT tube placement if needed with a unique guide system, beside to integrated fenestrated flap that protects from blockage with minimal increase in flow resistance. All these features of laryseal pro allow quick easy first time insertion success.

After approval of the Local Ethical Committee and obtaining an informed written consent from every patient, then patients will be categorized randomly into two equal groups using the computer allocation software to be put into opaque closed-envelopes: GL (n=27): Laryseal TM Pro. GA (n=27): Ambu Aura Gain.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55 years old
* ASA I& II
* Both sexes
* El-Ganzouri Airway Score < or =2

Exclusion Criteria:

* Active upper respiratory tract infections, pneumonia, COPD & exacerbated bronchial asthma.
* History of obstructive sleep apnea (OSA) or STOP Bang-Score > 4.
* Potentially full stomach (trauma, morbid obesity BMI> 35 Kg/m2, pregnancy, history of gastric regurgitation and heart burn).
* Esophageal reflux (hiatus hernia).
* Coagulation disorders.
* Patients with any cardiac conditions (IHD, RHD, decompensated heart failure and arrhythmia).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure (OLP) (cmH2O) | It will be measured at 5,15,30,45 and 60 minutes after successful SAD placement and effective ventilation.
  It is defined as the pressure at which leak starts. It will be calculated by the following steps : the adjustable pressure limit valve of the circle system is set at 60 cmH2O (airway pressures not allowed to exceed 40 cmH2O), the fixed fresh gas flow is set at 3 l.min-1, then the airway pressure is measured on the breathing system pressure gauge, so that leak pressure is considered as the achieved plateau airway pressure while the patient is apneic. At this stage an audible leak at the mouth (sound of gas escaping from mouth heard by listening close to patient's mouth) and stomach (sound of gas escaping into esophagus heard by auscultation over epigastrium) will be ascertained. To ensure safety, maximal allowable OLP will be fixed at 40 cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Reham Ali Abdelhaleem Abdelrahman, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Anesthesia, Surgical ICU, and Pain Management, Cairo, Egypt